CLINICAL TRIAL: NCT05231733
Title: A Phase 1, Open-label Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of an Anti-Claudin 18.2 Antibody SPX-101 in Patients With Advanced or Refractory Solid Tumors
Brief Title: Study of SPX-101 in Subjects With Advanced or Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Re-prioritized development strategy for this target
Sponsor: SparX Biotech(Jiangsu) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP21001
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPX-101 (Experimental): A total of up to 27 patients will be enrolled in this study. Subjects will receive SPX-101 by IV infusion in 60-minutes（±15 minutes）on Day 1 of the first cycle (3 weeks), and will be evaluated for DLTs in 3 weeks (DLT window). After the first cycle, subjects will continue the treatment at the assigned dose level.
  Interventions: Biological: SPX-101

INTERVENTIONS:
Biological: SPX-101 — Subjects will receive SPX-101 on Day 1 of the first cycle, and will be evaluated for DLTs in the following 3 weeks. After the first cycle, subjects will continue treatment at dosing intervals as determined by safety and PK results. All patients will continue treatment until disease progression, development of unacceptable toxicity, or until in the opinion of the investigator the patient is no longer benefiting from therapy, or at patient discretion (maximum duration: 2 years).

SUMMARY:
A Phase 1, Open-label Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of an anti-Claudin 18.2 Antibody SPX-101 in Patients with Advanced or Refractory Solid Tumors

DETAILED DESCRIPTION:
This is an open-label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics, and anti-tumor activity of various doses of SPX-101 in patients with advanced or refractory solid tumors.

This study will determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and select the recommended Phase2 dose (RP2D).

Up to five dose levels will be explored (1, 3, 9, 18, 30 mg/kg dose levels) depending on the number and intensity of observed toxicities.

A total of up to 27 patients will be enrolled in this study. Subjects will receive SPX-101 by IV infusion in 60-minutes（±15 minutes）on Day 1 of the first cycle (3 weeks), and will be evaluated for DLTs in 3 weeks (DLT window). After the first cycle, subjects will continue the treatment at the assigned dose level.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, refractory or recurrent disease of advanced solid tumors proven by histology, except for lung cancer.
* Subjects should not be eligible for curative surgery, and must have disease progression after treatment with available therapies that are known to confer clinical benefit or who are intolerant to or ineligible for standard treatment. There is no limit to the number of prior treatment regimens.
* Aged ≥18 years.
* Written informed consent.
* Eastern Cooperative Oncology Group performance status 0 to 2.
* Life expectancy >3 months.
* Adequate hepatic function; bilirubin <1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) <2.5 x ULN (5 x ULN if liver metastases was present).
* Adequate renal function; Cockcroft-Gault calculated creatine clearance (CrCl) or 24 hour urine CrCl ≥ 30 mL/min.
* Adequate hematological function: absolute neutrophil count ≥1.5 x 109/L; platelets ≥100 x 109/L; hemoglobin ≥9 g/dL (this can be post-transfusion).
* Women of childbearing potential (last menstruation <2 years prior to enrolment): negative blood serum pregnancy test (human chorionic gonadotropin) at screening phase and use of a highly effective method of contraception during the treatment phase and for 4 months after the last infusion of the study medication.
* Male patients whose sexual partners are women of childbearing potential must use condoms during the treatment phase and for 6 months after the last infusion of the study medication.
* The female partners of the male patients must also apply contraceptive methods.

Exclusion Criteria:

* Prior severe allergic reaction or intolerance to a monoclonal antibody, including humanized or chimeric antibodies. Prior severe allergic reaction or intolerance to any excipient in the formulations of the SPX-101 injection.
* Prior treatment with a claudin 18.2 Antibody
* Anti-tumor or radiotherapy treatment within 3 weeks of the start of study treatment (day 1 of cycle 1; a 2-week interval is allowed if palliative radiotherapy is given for peripheral bone metastases and the patient is recovered from acute toxicity).
* Use of other investigational agents or devices concurrently or within 4 weeks prior to study initiation (day 1 of cycle 1).
* Known human immunodeficiency virus infection or known symptomatic hepatitis (A, B, and/or C).
* Untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression.
* Clinically significant cardiac disease. History of myocardial infarction or hospitalization for congestive heart failure within 12 months of enrolment.
* Other clinically significant disease or comorbidity which may adversely affect the safe delivery of treatment within this study, including, but not limited to, any of the following: ongoing or active infection that required parenteral antibiotics, uncontrolled hypertension, clinically significant cardiac arrhythmia, or unstable angina pectoris.
* Psychiatric illness or social situations that would preclude study compliance.
* Pregnancy or breastfeeding.
* Gastric bleeding within the last 2 weeks; symptomatic peptic ulcer.
* Prior or current active autoimmune disease that required management with immunosuppression. This includes inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis, or other rheumatologic disease. Asthma and chronic obstructive pulmonary disease that did not require daily systemic corticosteroids is acceptable.
* Sinusoidal obstruction syndrome, formerly known as veno-occlusive disease, if present, should be stable or improving.
* Subject has Fridericia-corrected QT interval (QTcF) > 450 msec for males and > 470 msec for females on 12-lead electrocardiogram (ECG) at screening based on local testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD), and select the recommended Phase 2 dose (RP2D). | The analysis will extend through 28 days after the last administration of study drug.
  First-cycle dose limiting toxicities (DLTs). Adverse events as characterized by type, frequency, severity (as graded by NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.0), timing, seriousness and relationship to study therapy.
To determine the safety and tolerability of SPX-101 in patients with solid tumors | The analysis will extend through 28 days after the last administration of study drug.
  First-cycle dose limiting toxicities (DLTs). Adverse events as characterized by type, frequency, severity (as graded by NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.0), timing, seriousness and relationship to study therapy.

SECONDARY OUTCOMES:
To measure Area Under Curve (AUC) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To measure plasma clearance rate (CL) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To measure minimum concentration (Cmin) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To measure maximum concentration (Cmax) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To measure half-life (T1/2) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To measure apparent volume of distribution (Vd) | The analysis will extend through 28 days after the last administration of study drug.
  characterization of the pharmacokinetics (PK)
To assess Anti-Drug Antibody (ADA) | The analysis will extend through 28 days after the last administration of study drug.
  evaluating Immunogenicity
Objective response rate (ORR), as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) version1.1 | The analysis will extend through 28 days after the last administration of study drug.
  To evaluate antitumor efficacy
Disease control rate (DCR), as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) version1.1 | The analysis will extend through 28 days after the last administration of study drug.
  To evaluate antitumor efficacy
Duration of response (DOR), as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) version1.1 | The analysis will extend through 28 days after the last administration of study drug.
  To evaluate antitumor efficacy
Progression free survival (PFS), as assessed by Response Evaluation Criteria in Solid Tumor (RECIST) version1.1. | The analysis will extend through 28 days after the last administration of study drug.
  To evaluate antitumor efficacy

OTHER OUTCOMES:
To evaluate the capability of SPX-101 to induce immune effector-activity (ADCC) | The analysis will extend through 28 days after the last administration of study drug.
  Immune effector-activating capacity: Antibody-Dependent Cell-mediated Cytotoxicity (ADCC)
To evaluate the potential cytokine release induced by SPX-101, the activation of T cells including CD4+T and CD8+T cells will be analyzed | The analysis will extend through 28 days after the last administration of study drug.
  CD4+T and CD8+T cells

IPD SHARING:
Plan to Share IPD: No